CLINICAL TRIAL: NCT00068718
Title: Donor Lymphocyte Infusion for the Treatment of Malignancy After Hematopoietic Cell Transplantation Using Nonmyeloablative Conditioning - A Multi-center Trial
Brief Title: Donor Lymphocyte Infusion in Treating Patients With Persistent, Relapsed, or Progressing Cancer After Donor Hematopoietic Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1803.00; NCI-2010-00163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1803.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (DLI) (Experimental): Patients undergo unirradiated DLI over 15-30 minutes on day 0. Patients then undergo restaging on day 28 and may undergo a second DLI after at least 4 weeks if no significant GVHD develops and disease status worsens or after at least 8 weeks if disease status is unchanged and persistent donor T-cells are documented.
  Interventions: Biological: Therapeutic Allogeneic Lymphocytes

INTERVENTIONS:
Biological: Therapeutic Allogeneic Lymphocytes — Given IV
  Other Names: Allogeneic Lymphocytes

SUMMARY:
This phase I/II trial studies the side effects of donor lymphocyte infusion and to see how well it works in treating patients with persistent, relapsed (disease that has returned), or progressing cancer after donor hematopoietic cell transplantation. White blood cells from donors may be able to kill cancer cells in patients with cancer that has come back (recurrent) after a donor hematopoietic cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of donor lymphocyte infusion (DLI) as adoptive immunotherapy for persistent or relapsed malignant diseases in patients after related or unrelated nonmyeloablative transplantation.

SECONDARY OBJECTIVES:

I. To determine disease response, progression free and overall survival, chimerism, grade of graft-versus-host disease (GVHD), and infections.

OUTLINE:

Patients undergo unirradiated DLI over 15-30 minutes on day 0. Patients then undergo restaging on day 28 and may undergo a second DLI after at least 4 weeks if no significant GVHD develops and disease status worsens or after at least 8 weeks if disease status is unchanged and persistent donor T-cells are documented.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Only patients having received a preceding nonmyeloablative allogeneic transplantation with fludarabine/2 Gy total-body irradiation (TBI) - 4 Gy TBI or 2 Gy TBI - 4 Gy TBI conditioning from either a related or unrelated donor are eligible for this protocol
* Patients with persistent, relapsed or progressing malignancy after nonmyeloablative allogeneic transplantation; persistent disease will be defined as a failure to achieve a response as compared to baseline
* Patients with rapidly progressing malignancies (acute myeloid leukemia [AML], acute lymphocytic leukemia [ALL], blastic phase chronic myelogenous leukemia [CML-BC] intermediate-high-grade non-Hodgkin lymphoma [NHL], Hodgkin's lymphoma or aggressive multiple myeloma [MM]) should receive salvage chemotherapy or radiation before DLI according to the recommendation made in this protocol; any form of salvage chemotherapy should be discontinued no less than 3 weeks before DLI; therapy with Gleevec or interferon (IFN)-alpha should be discontinued prior to DLI; after salvage chemotherapy restaging is performed, patients with progressive disease and patients not meeting the inclusion criteria of the study after chemotherapy will be excluded from the study; patients are allowed to receive further doses of chemotherapy after DLI administration if they are scheduled for further DLI; after additional therapy the patients must be restaged and must again meet inclusion criteria to receive further DLI
* Patients must be able to tolerate a taper of systemic steroids to a dosage of less than or equal to 0.25 mg/kg/day; all other immunosuppressive therapy must have been discontinued for at least two weeks without significant flares in GVHD (i.e., increase of acute GVHD by one or more grades)
* Patients must have persistent donor cluster of differentiation (CD)3 cells (> 5% donor CD3 cells by a deoxyribonucleic acid [DNA]-based assay that compares the profile of amplified fragment length polymorphisms [ampFLP] [or fluorescent in situ hybridization (FISH) studies or variable number tandem repeat (VNTR)])
* DONOR: Alternatively to a fresh unmodified leukapheresis product, previously collected cryopreserved peripheral blood stem cells (PBSC) after mobilization with granulocyte colony-stimulating factor (G-CSF) or cryopreserved unmodified leukapheresis product from the original donor can be used; if cryopreserved product is not available, the DLI product must be from the original donor of hematopoietic cell transplantation
* DONOR: Original donor of hematopoietic cell transplantation
* DONOR: Donor must give consent to leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral or subclavian)
* DONOR: Donor must be medically fit to undergo the apheresis procedure (institutional guidelines for apheresis)

Exclusion Criteria:

* Current grade II to IV acute GVHD or extensive chronic GVHD
* Karnofsky score < 50%
* Lansky Play-Performance Score < 40 for pediatric patients
* DONOR: Donors who are not suitable for medical reasons to donate peripheral blood mononuclear cells (PBMC) by continuous centrifugation according to the criteria of the American Association of Blood Banks (AABB)
* DONOR: Pregnancy
* DONOR: Human immunodeficiency virus (HIV) or human T-lymphotrophic virus (HTLV) infection
* DONOR: Recent immunization may require a delay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (4):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- Universitaet Leipzig, Leipzig, Germany
- University of Torino, Torino, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (DLI)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 59.2 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 26
  Italy | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety of DLI Following a Non-myeloablative Transplant, Defined as Incidence of Grade IV Acute GVHD
Description: Percentage of Participants with Grade IV Acute GVHD
Time Frame: 100 days after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 5.7

2. Secondary Outcome: Incidence of Graft Rejection
Description: Percentage patients with graft rejection.
Time Frame: 100 days after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 5.7

3. Secondary Outcome: Incidence of Relapse/Progression
Description: CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever >38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  CMML, AML, ALL >30% BM blasts w/ deteriorating performance status, or worsening of anemia, neutropenia, or thrombocytopenia.
  CLL ≥1 of: Physical exam/imaging studies ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or number of plasmacytomas or lytic bone lesions.
Time Frame: 1 year after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 71.4

4. Secondary Outcome: Incidence of Grade II-IV GVHD in Patients Undergoing DLI Following a Non-myeloablative Transplant
Description: Percentage of Participants with II-IV Acute GVHD
Time Frame: 100 days after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 14.3

5. Secondary Outcome: Incidence of Infections in Patients Undergoing DLI Following a Non-myeloablative Transplant
Description: Percentage of Participants with infections.
Time Frame: 100 days after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 88.6

6. Secondary Outcome: Overall Survival
Description: Percentage patients surviving 1 year post-transplant.
Time Frame: 1 year after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 71.4

7. Secondary Outcome: Progression-free Survival
Description: Percentage of patients with progression-free survival
Time Frame: 1 year after DLI
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 35
percentage of participants | 28.6

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Treatment (DLI)
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (DLI) (N=35)
Blood bilirubin increased (Investigations) | 1 (1)
GVHD (Immune system disorders) | 3 (3)
Myocardial infaction (Cardiac disorders) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (DLI) (N=35)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
GVHD (Immune system disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (1)
Respiratory, thoracic, and mediastrinal disorders - Other (Unknown) (Renal and urinary disorders) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Metabolism and nutrition disorders - Other (Elevated tacrolimus level) (Metabolism and nutrition disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes